CLINICAL TRIAL: NCT01307007
Title: A Randomized, Controlled Study to Investigate the Safety and Explore the Mechanism of Hypophosphatemia With Intravenous Ferric Carboxymaltose (FCM) Versus Iron Dextran in Women With Iron Deficiency Secondary to Heavy Uterine Bleeding
Brief Title: Hypophosphatemia With Ferric Carboxymaltose Vs. Iron Dextran in Iron Deficiency Secondary to Heavy Uterine Bleeding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT08023
Record Dates: First submitted 2010-10-04; First posted 2011-03-02 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-01

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferric Carboxymaltose (FCM) (Experimental): 15 mg/kg up to a maximum of 1000 mg intravenous diluted in 250 cc normal saline solution administered over 15 minutes on Day 0
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Iron Dextran Injection (Active Comparator): Test dose of 25 mg administered over 5 minutes, if no reaction occurs then the remainder of the dose (15 mg/kg or 1000 mg including the test dose) will be administered as per investigator. The infusion must be given only when resuscitative techniques for the treatment of anaphylactic reactions are readily available.
  Interventions: Drug: Iron Dextran Injection

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM) — 15 mg/kg up to a maximum of 1000 mg intravenous diluted in 250 cc normal saline solution administered over 15 minutes on Day 0
  Other Names: Injectafer
  Arms: Ferric Carboxymaltose (FCM)
Drug: Iron Dextran Injection — Test dose of 25 mg administered over 5 minutes, if no reaction occurs then the remainder of the dose (15 mg/kg or 1000 mg including the test dose) will be administered as per investigator. The infusion must be given only when resuscitative techniques for the treatment of anaphylactic reactions are readily available.
  Other Names: Dexferrum and INFeD
  Arms: Iron Dextran Injection

SUMMARY:
The primary objective of this study is to assess the safety of an investigational intravenous iron (ferric carboxymaltose [FCM]) or an equal dose of iron dextran and explore the mechanism of hypophosphatemia following administration of FCM or that of an equal dose of iron dextran when treating women with iron deficiency anemia due to heavy uterine bleeding (HUB).

DETAILED DESCRIPTION:
To assess the safety of an investigational intravenous iron (ferric carboxymaltose [FCM]) or an equal dose of iron dextran and explore the mechanism of hypophosphatemia following administration of FCM or that of an equal dose of iron dextran when treating women with iron deficiency anemia due to heavy uterine bleeding (HUB).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects > or = to 18 years of age
* History of Heavy Uterine Bleeding within the past 6 months
* Screening visit central laboratory Hgb < 12 g/dL
* Screening Visit ferritin < or = to 100 ng/mL or < or = to 300 when transferrin saturation (TSAT) is < or = to 30%
* Demonstrate the ability to understand the requirements of the study, willingness to abide by study restrictions and to return for the required assessments

Exclusion Criteria:

* Known hypersensitivity reaction to any component of ferric carboxymaltose or iron dextran
* Previously randomized in a clinical study of ferric carboxymaltose
* Requires dialysis for treatment of chronic kidney disease
* Chronic kidney disease, marked by estimated glomerular filtration rate < 60 ml/min/1.73m squared
* Previous kidney transplant
* History of primary hypophosphatemic disorder
* Hypophosphatemia < 2.6 mg/dl
* No evidence of iron deficiency
* During the 10 day period prior to screening has been treated with intravenous iron
* During the 30 day period prior to screening or during the study period has or will be treated with erythropoiesis stimulating agents (ESA) in a regimen that is off label
* During the 30 day period prior to screening or during the study period has or will be treated with a red blood cell transfusion, radiotherapy and/or chemotherapy
* During the 30 day period prior to screening or during the study period has or will require a surgical procedure that necessitates general anesthesia
* Any non-viral infection
* Aspartate aminotransferase (AST) or Alanine Aminotransferase (ALT) at screening, as determined by central labs, greater than 1.5 times the upper limit of normal
* Known positive hepatitis with evidence of active disease
* Received an investigational drug within 30 days of screening
* Alcohol or drug abuse within the past 6 months
* Hemochromatosis or other iron storage disorders
* Malignancy history within the past 5 years other than basal or squamous cell skin cancer
* Any other laboratory abnormality, medical condition or psychiatric disorders which in the opinion of the investigator would put the subject's disease management at risk or may result in the subject being unable to comply with study requirements
* Pregnant or sexually-active female subjects who are of childbearing potential and who are not willing to use an acceptable form of contraception
* Untreated primary hyperparathyroidism
* Untreated gastrointestinal malabsorption (e.g., sprue)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Falone, MD, Study Director — American Regent, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wolf M, Koch TA, Bregman DB. Effects of iron deficiency anemia and its treatment on fibroblast growth factor 23 and phosphate homeostasis in women. J Bone Miner Res. 2013 Aug;28(8):1793-803. doi: 10.1002/jbmr.1923. PMID 23505057
- See also: FGF23; IRON; PHOSPHATE; PTH; VITAMIN D — https://www.ncbi.nlm.nih.gov/pubmed/23505057

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and medical clinics
Pre-assignment Details: In the FCM group, reasons for discontinuation prior to dosing included lost to follow-up (5 subjects), subject request (2 subjects), and selection criteria/study compliance (2 subjects). In the iron dextran group, reasons for discontinuation prior to dosing included subject request (4 subjects) and lost to follow-up (1 subject).
Groups:
- Ferric Carboxymaltose (FCM): Ferric Carboxymaltose (FCM) : 15 mg/kg up to a maximum of 1000 mg intravenous diluted in 250 cc normal saline solution administered over 15 minutes on Day 0
- Iron Dextran Injection: Iron Dextran Injection : Test dose of 25 mg administered over 5 minutes, if no reaction occurs then the remainder of the dose (15 mg/kg or 1000 mg including the test dose) will be administered as per investigator. The infusion must be given only when resuscitative techniques for the treatment of anaphylactic reactions are readily available.
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Dextran Injection
Started | 25 | 30
Completed | 25 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Dextran Injection | Total
Number analyzed (Participants) | 25 | 30 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 30 | 55
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (10.26) | 33.7 (10.72) | 35.1 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 55
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 30 | 55

OUTCOME MEASURES:

1. Primary Outcome: Changes in Blood Markers
Description: Changes in blood markers of phosphate
Time Frame: Day 35
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Dextran Injection
Number analyzed (Participants) | 21 | 26
mg/dL | -.38 (.878) | -.08 (.633)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Dextran Injection
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/30
Other Adverse Events (participants affected / at risk) | 12/25 | 14/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=25) | Iron Dextran Injection (N=30)
Nausea (Gastrointestinal disorders) | 1 | 2
Edema peripheral (General disorders) | 0 | 2
Hypersensitivity (Immune system disorders) | 2 | 1
Sinusitis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 8 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days